CLINICAL TRIAL: NCT04164758
Title: A Pilot Randomized, Double-blind, Placebo-controlled Study to Evaluate Safety and Daytime Sedation in Subjects With Parkinson's Disease With Neuropsychiatric Symptoms Treated With Pimavanserin or Low-Dose Quetiapine
Brief Title: Study to Evaluate Safety and Daytime Sedation in Subjects With Parkinson's Disease With Neuropsychiatric Symptoms Treated With Pimavanserin or Low-Dose Quetiapine
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study enrollment impacted by COVID-19 pandemic and Sponsor terminated for business reasons
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-056
Record Dates: First submitted 2019-11-13; First posted 2019-11-15 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — pimavanserin; Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Drug - pimavanserin (Experimental): Pimavanserin 34 mg provided as 2 x 17 mg encapsulated tablets
  Interventions: Drug: Pimavanserin
- Placebo (Placebo Comparator): Placebo encapsulated tablet
  Interventions: Other: Placebo
- Quetiapine (Active Comparator): Immediate release Quetiapine encapsulated tablets
  Interventions: Drug: Quetiapine

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg (provided as 2×17 mg encapsulated tablets) administered orally as a single dose once daily
  Arms: Drug - pimavanserin
Other: Placebo — Placebo (provided as 2 × placebo encapsulated tablets) administered orally as a single dose once daily
  Arms: Placebo
Drug: Quetiapine — Quetiapine 25 mg (provided as 1×25 mg quetiapine encapsulated tablet and 1 × placebo encapsulated tablet), OR 50 mg (provided as 2×25 mg quetiapine encapsulated tablets), OR 100 mg (provided as 2×50 mg quetiapine encapsulated tablets) administered orally as a single dose once daily
  Arms: Quetiapine

SUMMARY:
This is a pilot study to explore the effects of pimavanserin and low-dose quetiapine in subjects with Parkinson's disease with neuropsychiatric symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 50 to 85 years of age, inclusive
2. Able to understand the protocol requirements and provide written informed consent
3. Able to complete questions on a handheld device / tablet, is willing to wear an actigraph and can be reliably rated on assessment scales
4. Able to designate an 'informant' (relative, housemate, friend) who can provide information about the subject's well being and attend clinic visits with the subject
5. Is able to swallow the test capsule without difficulty during the Screening visit
6. Has a Mini-Mental State Examination (MMSE) score ≥19
7. Has a diagnosis of idiopathic Parkinson's disease, without any other known or suspected cause of parkinsonism. Initial diagnosis of PD must have been made more than 1 year prior to Screening.
8. Has non-motor neuropsychiatric symptoms severe enough to warrant treatment with an antipsychotic agent based on investigator judgement and CGI-S score
9. If the subject is on anti-Parkinsonian medication, they must be on a stable regimen for 1 month prior to Baseline and not planning (at the time of the Baseline visit) to make a major change in dose(s)
10. If the subject is female, she must not be pregnant or breastfeeding. She must also be of non-childbearing potential or must agree to use a clinically acceptable method of contraception or be abstinent for at least 1 month prior to the Baseline visit, during the study, and 41 days following completion of double-blind treatment.

Exclusion Criteria:

1. Has atypical parkinsonism or secondary parkinsonism variants such as tardive or medication induced parkinsonism
2. Is in hospice, is receiving end-of-life palliative care, or is bedridden or confined to a wheelchair
3. Has neuropsychiatric symptoms that are primarily attributable to current delirium or substance abuse
4. Has current evidence of an unstable neurological, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical or psychiatric disorder, including cancer or malignancies that, in the judgment of the Investigator, would jeopardize the safe participation of the subject in the study or significantly interfere with the conduct or interpretation of the study
5. Has a known personal or family history of long QT syndrome or family history of sudden cardiac death
6. Has orthostatic hypotension as judged by the investigator and medical monitor
7. Is judged by the Investigator or the Medical Monitor to be inappropriate for the study for any reason, including if the subject is judged to be a danger to self or others

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all pre-specified entry criteria).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-23 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Tucson Neuroscience Research, Tucson, Arizona
  - Sutter Institute for Medical Research, Sacramento, California
  - Galiz Research, Hialeah, Florida
  - Charter Research, LLC, Lady Lake, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Charter Research, LLC, Winter Park, Florida
  - Meridian Clinical Research, Savannah, Georgia
  - Hawaii Pacific Neuroscience, LLC., Honolulu, Hawaii
  - University of lowa Hospital and Clinics, Iowa City, Iowa
  - SRI International, Plymouth, Michigan
  - Bio Behavioral Health, Toms River, New Jersey
  - M3 Wake Research, Inc., Raleigh, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - Prisma Health-Upstate, Greenville, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in patients aged 50-85 years with a diagnosis of idiopathic Parkinson's disease (PD) with a minimum duration of >1 year at screening and with no other known or suspected cause of parkinsonism.
Pre-assignment Details: During the screening period, patients were assessed for study eligibility, and prohibited medications were discontinued when medically appropriate.
Groups:
- Placebo: Two encapsulated placebo tablets, taken once daily
- Quetiapine: Quetiapine starting dose 25 mg once daily (provided as 1 × 25 mg quetiapine immediate release encapsulated tablet plus 1 placebo encapsulated tablet), with the possibility to increase the dose to 50 mg (2 × 25 mg quetiapine immediate release encapsulated tablets) or 100 mg (2 × 50 mg quetiapine immediate release encapsulated tablets) taken once daily, based on clinical response.
- Pimavanserin 34 mg: Pimavanserin provided as 2 × 17 mg encapsulated tablets, taken once daily
Period: Overall Study
Arm/Group | Placebo | Quetiapine | Pimavanserin 34 mg
Started | 4 | 4 | 3
Completed | 3 | 3 | 3
Not Completed | 1 | 1 | 0
Not completed — COVID-19 withdrawal of consent | 1 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Analysis set, i.e. all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Quetiapine | Pimavanserin 34 mg | Total
Number analyzed (Participants) | 4 | 4 | 3 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.8 (5.74) | 68.0 (8.49) | 62.0 (3.00) | 67.0 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 4
  Male | 1 | 4 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 4 | 3 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 3 | 11

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Assess the safety and tolerability of pimavanserin in patients with PD in terms of treatment-emergent adverse events.
Time Frame: 4-week treatment duration, plus 30 days treatment-free safety follow-up
Population: Safety Analysis set, i.e. all patients who had received at least one dose of study medication
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Quetiapine | Pimavanserin 34 mg
Number analyzed (Participants) | 4 | 4 | 3
Participants | 1 | 3 | 1

ADVERSE EVENTS:
Time Frame: 4-week treatment duration, plus 30 days treatment-free safety follow-up
Arm/Group | Placebo | Quetiapine | Pimavanserin 34 mg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 1/4 | 3/4 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | Quetiapine (N=4) | Pimavanserin 34 mg (N=3)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
In March 2020, recruitment of new patients was paused due to the emerging coronavirus disease 2019 (COVID-19) pandemic. It was restarted in Jun 2020 and paused again in Aug 2020. Subsequently, no further patients were enrolled. On 24 Sep 2020, the sponsor decided to permanently stop the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator may publish the study results, relative to their own patients, only after review, comment and approval by the sponsor. No publication of confidential information shall be made without the sponsor's prior written consent. At least 60 days prior to submitting a manuscript or prior to any public presentation, a copy of the manuscript or presentation will be provided to the Sponsor for review and comment. The sponsor has 60 days to review and comment.

DOCUMENTS (2):
  • Study Protocol (2020-01-31): https://cdn.clinicaltrials.gov/large-docs/58/NCT04164758/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT04164758/SAP_001.pdf